CLINICAL TRIAL: NCT06244108
Title: The Effect of Occupational Therapy Home Programs on Sensory Processing and Feeding Problems in Children With Down Syndrome: A Randomised Controlled Trial
Brief Title: Occupational Therapy Home Programs in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zengin0001
Record Dates: First submitted 2024-01-10; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Down Syndrome; Occupational Therapy; Feeding Problem
Keywords: Down Syndrome; Occupational Therapy; Home Program; Sensory Function; Randomized; Control Trial
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Two groups. Intervention and control groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTHP Group (Intervention Group) (Experimental): Children with Down syndrome will undergo an 8-week occupational therapy home program (OTHP). Evaluations will be conducted at the beginning and end of the intervention, and the results will be compared.
  Interventions: Other: Occupational therapy home program
- None OTHP Group (Control group) (No Intervention): The control group (non-OTHP) will not receive occupational therapy home program, even if they have Down syndrome. Evaluations will be conducted at 8-week intervals, with the first and last evaluations being compared.

INTERVENTIONS:
Other: Occupational therapy home program — After evaluating the children, an occupational therapy home intervention program will be developed for each child. The program will be monitored through telephone and computer interviews, as well as video, photo, and audio recordings. The interventions in this study were selected based on successful occupational therapy home programs for children with disabilities. The program consists of five steps.
  Step 1 is to establish collaborative relationships with parents. Step 2 is to determine the most appropriate goals for the child and their family. Step 3 involves selecting the most suitable therapeutic activities to achieve these goals. Step 4 is to educate and support parents in performing these therapeutic activities. Finally, Step 5 involves measuring the results and providing feedback.
  Arms: OTHP Group (Intervention Group)

SUMMARY:
Children with Down Syndrome frequently encounter difficulties with sensory functions and feeding, such as oral sensory processing issues and developmental disorders. The aim of this study was to examine the effects of an Occupational Therapy Home Program on the sensory functions and feeding issues of children with Down Syndrome.

DETAILED DESCRIPTION:
Although there are studies that investigate nutritional issues in children with Down syndrome, no well-structured, high-evidence, and individual-centered studies have been found. The literature assumes a relationship between the sensory functions and nutritional status of children with Down syndrome. Therefore, further studies are needed to develop intervention programs to prevent sensory processing and nutritional problems.

This study aims to evaluate the effectiveness of occupational therapy home programs in improving sensory functions and feeding problems in children with Down syndrome. The study focuses on evidence-based practices to assess the impact of these programs compared to not providing them.

The study will be conducted with children diagnosed with Down Syndrome who have applied to the Pediatrics Unit of the Department of Occupational Therapy at Hacettepe University Faculty of Health Sciences.

The study comprises pre-evaluation, final evaluation, and intervention stages. Following the initial evaluation, an occupational therapy home intervention program will be implemented for the children before and after each meal, seven days a week, for eight weeks. Evaluations will be repeated after the eight-week period.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 3-10
* Having Down Syndrome
* Families agree to participate in the study

Exclusion Criteria:

* Having previously received sensory integration and/or occupational therapy treatment
* Having a secondary diagnosis other than Down Syndrome (Mental Retardation, etc.)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Sensory Profile | 8 weeks
  The Sensory Profile developed by Winnie Dunn was used to evaluate sensory processing skills in Turkish. This assessment is suitable for children aged three to ten. The test is completed by an occupational therapist, accompanied by the person who has the most contact with the child in their daily life. Each item is scored on a Likert scale from 1 to 5. The Sensory Profile consists of three parts: sensory processing, modulation, and behavioral-emotional responses. Each part has 14 parameters. The score indicates the level of sensitivity, with lower scores indicating hypersensitivity, higher scores indicating hyposensitivity, and middle values indicating typical performance.
Screen Tool of Feeding Problems (STEP) | 8 weeks
  The study used the Systematic Tool for Evaluating Progress (STEP) to identify feeding challenges and problematic feeding behaviours experienced by individuals with Down Syndrome (DS). STEP includes questions for parents or personnel who have worked with the individual for the last six months, asking about any abnormal behaviours observed in the last month. The survey consists of 23 items, each addressing a specific nutritional issue. The aforementioned issues are categorized into five subgroups: aspiration risk, food selectivity, feeding skills, behavioural problems related to food rejection, and behavioural problems related to nutrition. The study used the Systematic Tool for Evaluating Progress (STEP) to identify feeding challenges and problematic feeding behaviours experienced by individuals with Down Syndrome (DS). An increase in the score suggests an increase in nutritional problems.
Demographic Form | 8 weeks
  The form completed by the child's primary caregiver includes information such as the child's age, gender, number of siblings, and the marital status of both parents.
A meal time | 8 weeks
  The study recorded the child's average meal time as reported by their parents during the first and last evaluations. The event was documented in the minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gökçen Akyürek, Assoc. Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study's completion is anticipated to result in a scientific article that will contribute to evidence-based practices.